CLINICAL TRIAL: NCT05874375
Title: Safety and Performance of UCon for Management of Non-Neurogenic OAB in Males - An Early Feasibility Study
Brief Title: UCon Treatment of Overactive Bladder (OAB) in Males
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: InnoCon Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NL_FEAS_01
Record Dates: First submitted 2023-05-01; First posted 2023-05-24 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Urinary Incontinence; Urge Incontinence; Nocturia; Urinary Frequency More Than Once at Night; Urinary Incontinence, Urge; Incontinence, Nighttime Urinary
Keywords: Urinary Incontinence; Urge incontinence; Neurostimulation; Dorsal Genital Nerve; Nocturia
MeSH Terms: conditions — Urinary Incontinence; Urinary Incontinence, Urge; Nocturia; Nocturnal Enuresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Urge and Time limited) (Other): The participant self-administer electrical stimulation to the dorsal genital nerve (DGN) using UCon with a stimulation mode that is activated for 60 seconds by the participant when he experience urgency (urge stimulation).The urge stimulation can be activated repeatedly during the day as the participant wears the device from morning to evening at home for 14 days. Following a stimulation wash-out period (14 days), the participants then stimulates with UCon for another 14 days using the time limited stimulation mode.
  Interventions: Device: Urge stimulation; Device: Time limited stimulation
- Group B (Time limited and Urge) (Other): The participant self-administer electrical stimulation to the dorsal genital nerve (DGN) using UCon with a stimulation mode that is activated for 30 minutes once a day, at a time that is convenient for the participant. The participant uses the device at home for 14 days. Following a stimulation wash-out period (14 days), the participant then stimulates with UCon for another 14 days using the urge stimulation mode.
  Interventions: Device: Urge stimulation; Device: Time limited stimulation

INTERVENTIONS:
Device: Urge stimulation — Participants will receive stimulation for 60 seconds, when they feel an urgency.
  Other Names: DGN stimulation; Neurostimulation
Device: Time limited stimulation — Participant will receive the stimulation as provided in time limited sessions (Range: 15 min - continuous), whenever it suits the participant during the day.
  Other Names: DGN stimulation; Neurostimulation

SUMMARY:
UCon is a medical device for treatment of the symptoms of OAB and fecal incontinence (FI). It electrically stimulates the DGN through the skin to obtain modulated behaviour of the bladder musculature e.g., suppress undesired bladder activity to relieve the symptoms of the patient. This clinical investigation is a randomized, cross-over, single-site, prospective, early feasibility study, which is used to evaluate Ucon with respect to its initial clinical safety and device performance in a small number of males with OAB.

DETAILED DESCRIPTION:
The purpose of the current investigation is to obtain information about the type of stimulation that Ucon provide (time limited vs. urge stimulation), would be the most effective and feasible for the treatment of non-neurogenic OAB symptoms in males.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥ 18 years of age.
2. Subject is male.
3. Subject is diagnosed with OAB
4. Subject is able to communicate, provide feedback, understand and follow instructions during the course of the investigation.

Exclusion Criteria:

1. Subject is medically unstable (acute illness or complications of a chronic condition that might affect the subject's participation in the investigation).
2. Subject has a Post Void Residual (PVR) of more than 100 ml or a Bladder Voiding Efficiency (BVE) of less than 75% (measured by uroflowmetry as the ratio of voided volume (VV) and total bladder capacity (VV+PVR)).
3. Subject has an active infection in the genital area incl. skin infections and urinary tract infection.
4. Subject has had botulinum toxin (BOTOX) treatment in the pelvic region within 6 months.
5. Subject has used antimuscarinics or β3 agonists within 14 days weeks*.
6. Subject has an implanted pacemaker, implantable drug pump or other active medical device (any medical device that uses electrical energy or other source of power to make it function).
7. Subject is enrolled or planning to enrol in another clinical investigation or was enrolled in an investigational drug study or medical device investigation within four weeks to enrolment.
8. Subject has neuropathy to a degree that is presumed to diminish the effect of the electrical stimulation.
9. Subject has a history of cancer in the pelvic region, are currently receiving cancer treatment, or has radiation-induced damage to the pelvic region.
10. Subject has addictive behaviour defined as abuse of alcohol, cannabis, opioids, or other intoxicating drugs.
11. Subject does not speak and understand Dutch.

    * If a subject is currently being treated with antimuscarinics or β3 agonists, he is allowed to be included in the investigation, however, a washout period of 14 days is required before baseline can be established.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-10-12 (Actual); Primary Completion 2026-06-12 (Estimated); Study Completion 2026-06-12 (Estimated)

PRIMARY OUTCOMES:
PRIMARY SAFETY: To evaluate adverse events [initial safety] of UCon for treatment of OAB symptoms in a home setting. | After 44 days (end of study)
  Characterization of adverse events and anticipated adverse device effects associated with the use of UCon during the investigational period.
PRIMARY PERFORMANCE: To evaluate the ratio of treatment change [performance] of OAB symptoms using UCon in a home setting | Change from baseline at 14 days, 30 days and 44 days (study end)
  Ratio of subjects with at least 50% change in their OAB symptoms from baseline. Participants shall complete a 3-day bladder diary to report their symptoms.
  The symptoms related to OAB:
  * Urinary urgency is measured by number of urgency episodes/day.
  * Urinary frequency is measured by number of voidings/day.
  * Urgency urinary incontinence is measured by number of leaks preceded by urgency/day.
  * Nocturia is measured by number of voidings/night.

SECONDARY OUTCOMES:
SECONDARY SAFETY: To identify the number of subjects experiencing adverse events associated with the use of UCon during the investigational period. | After 44 days (end of study)
  Number of subjects experiencing adverse events and anticipated adverse device effects. Subjects will report on any experience associated with the use of UCon.
SECONDARY SAFETY: To evaluate the severity of adverse events associated with the use of UCon during the investigational period. | After 44 days (study end)
  Severity of adverse events and anticipated adverse device effects.The severity will be evaluated from the subjects' report on any experience associated with the use of UCon.
SECONDARY PERFORMANCE: To evaluate whether subjects using UCon experience a change in their quality of life. | Change from baseline at 14 days and 44 days (end of study)
  Ratio of subjects with a change in their OAB quality of life measures as assessed by specific QoL questionnaires related to OAB condition (ICIQ-OAB, AOBq). An overall score with greater values indicates a worse symptom outcome.
SECONDARY PERFORMANCE: To evaluate whether subjects using UCon experience a change in their treatment outcome (i.e. symptoms) after therapy. | Change from baseline at 14 days and 44 days (end of study)
  Ratio of subjects with a change in their treatment outcome (i.e. symptoms) assessed by the 7-point Patient Global Impression of Improvement (PGI-I) scale. Higher scores indicates a worse treatment outcome.
SECONDARY PERFORMANCE: To evaluate the device and treatment acceptability of UCon. | After 44 days (study end)
  Ratio of subjects that accept UCon and DGN stimulation as assessed by a satisfaction survey recorded after each stimulation period.

CONTACTS AND LOCATIONS:
Overall Officials: John Heesakkers, MD, Principal Investigator — Maastricht UMC+, P. Debyelaan 25, 6229 HX Maastricht, The Netherlands
Locations (1):
- Maastricht University Medical Center+, Maastricht, Netherlands